CLINICAL TRIAL: NCT05060757
Title: Microbiome Test for the Detection of Colorectal Polyps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biotax Labs LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Biotax_001
Record Dates: First submitted 2021-09-19; First posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Colon Polyp
Keywords: Colonoscopy; microbiome; colon polyp
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- colonoscopy (Experimental): Participants will be patients undergoing colonoscopy
  Interventions: Diagnostic Test: biotax

INTERVENTIONS:
Diagnostic Test: biotax — patients who are scheduled to undergo colonoscopy will be asked to participate and give a stool sample

SUMMARY:
The main goal of this trial is to validate a new method for colorectal polyp screening based on stool microbiome signatures. 600 Individuals who are scheduled / planned to undergo a colonoscopy will be recruited for this study and a stool sample and an optional saliva sample will be collected.

Analyze process will be conducted on the microbiome of the samples given.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second cause of cancer death in the US. The pathogenesis of CRC is complex, involving a progressive transition of the healthy colonic mucosa to pre-cancerous polyps, and eventually to CRC. One of the factors that are proposed to cause this 'adenoma-carcinoma sequence' is the dysbiosis of the gut microbiome.

The gut microbiota has been identified as a potential screening biomarker for CRC, since studies have reported specific bacterial taxa and/ or microbial signatures as important factors in the etiology of CRC.

Hypothesis:

comprehensive and cutting-edge metagenomic analysis of the fecal microbiome of individuals with colonic polyps vs. patients without polyps will identify microbial signatures associated with colonic polyps and will define these microbial signatures as biomarkers and risk factors for CRC.

method:

* Collect data (anthropometric, demographic, dietary, lifestyle habits, medical and family history) and stool & optional Saliva sample for microbiome analysis from a cohort of 600 colonoscopies screened individuals.
* Analyze this data with an aim to utilize advanced artificial intelligence and machine-learning techniques to classified microbiome signatures, which are correlated to colonoscopy (and to histological) results.
* Blinded Validation - A sub-cohort of 300 individuals (who are part of the 600 individuals) that were not used to classify the biomarkers signatures will be used to validate the diagnosis model.

Data analysis:

The stool and optional Saliva samples will be sent to metagenomic sequencing, thereby generating FASTQ libraries of the reads found in the stool & saliva samples. These files will be analyzed by the BiotaX diagnostics platform.

No Human DNA analysis will take place at this clinical study. Only a microbial analysis will take place.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females.
2. Age: 45-70 years, inclusive.
3. Patients without any incapacitating systemic disease
4. Able to comprehend and provide informed consent.
5. Patients who are scheduled / planned to undergo a colonoscopy, preferably: participants who are undergoing a colonoscopy as a diagnostic surveillance.

Exclusion Criteria:

1. Subject has a history of colorectal cancer (CRC)
2. Subject has a diagnosis or medical history of any of the following conditions:

   * Familial adenomatous polyposis (also referred to as "FAP", including attenuated FAP and Gardner's syndrome)
   * Hereditary non-polyposis CRC syndrome (also referred to as "HNPCC" or "Lynch Syndrome")
3. Subject has a diagnosis or personal history of inflammatory bowel disease (IBD), including chronic ulcerative colitis or Crohn's disease.
4. Patients with incapacitating systemic disease
5. Any use of antibiotics within one months prior to colonoscopy.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-07-27 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
diagnose existence of colon polyps | year
  To determine whether fecal metagenomics microbial signatures can significantly predict adenoma\ sessile serrated polyps (SSP) existence in patients and serve as diagnostic biomarkers.

SECONDARY OUTCOMES:
diagnose sub types of colon polyps | year
  To determine whether fecal metagenomics microbial signatures can significantly identify between the following subgroups: non-polyp group, Hyperplastic polyps, adenomas - <5 mm, 6-10mm polyp group and >10mm polyp group.
Saliva microbiome vs stool microbiome | year
  To determine if Saliva microbiome sample can provide indication same as Stool microbiome sample.

CONTACTS AND LOCATIONS:
Overall Officials: Zohar Levi, MD, Principal Investigator — Assuta Medical Center; Erez Hasnis, MD, Principal Investigator — Rambam Health Care Campus
Locations (2):
- Israel (2):
  - Rambam Medical Center, Haifa
  - Assuta Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dadkhah E, Sikaroodi M, Korman L, Hardi R, Baybick J, Hanzel D, Kuehn G, Kuehn T, Gillevet PM. Gut microbiome identifies risk for colorectal polyps. BMJ Open Gastroenterol. 2019 May 27;6(1):e000297. doi: 10.1136/bmjgast-2019-000297. eCollection 2019. PMID 31275588
- [Background] Garrett WS. The gut microbiota and colon cancer. Science. 2019 Jun 21;364(6446):1133-1135. doi: 10.1126/science.aaw2367. No abstract available. PMID 31221845
- [Background] Thomas AM, Manghi P, Asnicar F, Pasolli E, Armanini F, Zolfo M, Beghini F, Manara S, Karcher N, Pozzi C, Gandini S, Serrano D, Tarallo S, Francavilla A, Gallo G, Trompetto M, Ferrero G, Mizutani S, Shiroma H, Shiba S, Shibata T, Yachida S, Yamada T, Wirbel J, Schrotz-King P, Ulrich CM, Brenner H, Arumugam M, Bork P, Zeller G, Cordero F, Dias-Neto E, Setubal JC, Tett A, Pardini B, Rescigno M, Waldron L, Naccarati A, Segata N. Author Correction: Metagenomic analysis of colorectal cancer datasets identifies cross-cohort microbial diagnostic signatures and a link with choline degradation. Nat Med. 2019 Dec;25(12):1948. doi: 10.1038/s41591-019-0663-4. PMID 31664237
- See also: colorectal cancer statistics — https://www.cancer.org/cancer/colon-rectal-cancer/about/key-statistics.html